CLINICAL TRIAL: NCT06411457
Title: Single-arm, Multi-center Phase II Clinical Study of SHR-A1811 in Combination With Adebrelimab for the Treatment of HER2 Low-expressing Metastatic Breast Cancer
Brief Title: SHR-A1811 in Combination With Adebrelimab for the Treatment of HER2 Low-expressing Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, QIAO LI, Clinical Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4483
Record Dates: First submitted 2024-05-04; First posted 2024-05-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811+Adebrelimab (Experimental): Assess the efficacy and safety of the SHR-A1811 in combination with Adebrelimab regimen in HER2 low-expressing metastatic breast cancer
  Interventions: Drug: SHR-A1811+Adebrelimab

INTERVENTIONS:
Drug: SHR-A1811+Adebrelimab — Assess the efficacy and safety of the SHR-A1811 in combination with Adebrelimab regimen in HER2 low-expressing metastatic breast cancer SHR-A1811 : 6.4mg/kg , q3w，d1, ivgtt Adebrelimab : 1200mg, q3w，d1, ivgtt

SUMMARY:
To evaluate the efficacy and safety of the SHR-A1811 in combination with Adebrelimab regimen in HER2 low-expressing metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years; ER/PgR expression ≤10% and low HER2 expression (IHC 1+, or IHC 2+ and ISH-); Advanced breast cancer patients; Prior treatment with ≥1 line of therapy for localized recurrence or metastatic disease; At least one prior treatment with taxane or anthracycline therapy; Allowed to receive immunotherapy during neoadjuvant or adjuvant stages; Measurable lesions according to RECIST 1.1 standards; ECOG PS score: 0-1; Voluntary participation with good compliance; Negative pregnancy test result, childbearing-age participants commit to effective contraception from the study start to 6 months after the last dose; Adequate organ function; Blood routine: ANC ≥1.5×109/L, PLT≥70×109/L, HGB ≥90g/L; Liver function: TBIL ≤1.5×ULN, ALT and AST ≤3×ULN, serum albumin ≥28 g/L, ALP ≤5×ULN; Stable liver function for at least 1 week after routine liver protection treatment, as assessed by the investigator, is eligible for inclusion; Renal function: Cr ≤1.5×ULN, or CrCl ≥50 mL/min (using standard Cockcroft-Gault formula); Coagulation function: INR ≤1.5/PT ≤1.5×ULN, aPTT ≤1.5×ULN; Left ventricular ejection fraction ≥50%

Exclusion Criteria:

- Active central nervous system metastases or carcinomatous meningitis (stable brain metastasis patients are allowed to participate); Prior treatment with anti-HER2 ADC drugs; Active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; Patients with vitiligo; Childhood asthma completely resolved in adulthood without any intervention can be included, but asthma requiring bronchodilators for medical intervention in adulthood cannot be included); Patients using immunosuppressants or systemic steroid therapy for immunosuppressive purposes (dose>10mg/day prednisone or equivalent) in the 2 weeks before inclusion; Patients with other malignant tumors in the past or simultaneously; Grade ≥4 adverse reactions after ADC drug treatment, grade ≥3 immune-related adverse reactions; Known allergy to drug components used; Patients with known interstitial pneumonia; Poorly controlled clinical heart symptoms or diseases, such as: (1) NYHA class 2 or above heart failure; (2) unstable angina; (3) myocardial infarction within the past year; (4) patients with clinically significant ventricular or supraventricular arrhythmias requiring treatment or intervention; Active infection or unexplained fever >38.5°C during the screening period or before the first dose of study medication, depending on the investigator's judgment, patients with fever due to tumor can be included; Not receiving live vaccines within less than 4 weeks before or during the study; Patients known to have a history of psychiatric drug abuse, alcoholism, or drug addiction; Factors that may lead to the premature termination of the study judged by the investigator, such as other serious diseases (including mental illness) requiring concomitant treatment, severe laboratory abnormalities, family or social factors affecting patient safety, data and sample collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-16 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
ORR | ORR date will be assessed evey 6 weeks starting from the randomization date until first documented progression or date of death from any cause whichever came first assessed up to 3 years
  Overall response rate

SECONDARY OUTCOMES:
3-month PFS | 3-month progression-free survival rate will be assessed evey 6 weeks starting from the randomization date until first documented progression or date of death from any cause which ever came first assessed up to 3 month.
  progression-free survival rate at 3 month
PFS | progression date will be assessed evey 6 weeks starting from the randomization date until first documented progression or date of death from any cause whichever came first assessed up to 3 years
  Progression-free survival
Clinical benefit rate (CBR) | CBR will be assessed evey 6 weeks starting from the randomization date until first documented progression or date of death from any cause whichever came first assessed up to 3 years
Safety endpoints | Safety date will be assessed evey 6 weeks starting from the randomization date until first documented progression or date of death from any cause whichever came first assessed up to 3 years
  including incidence of adverse events (AE), serious adverse events (SAE), and immune-related adverse events (irAE)

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Li, M.D., Principal Investigator — National Cancer Center/Cancer Hospital
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No